CLINICAL TRIAL: NCT06224569
Title: Quantifying the Effects of Daily Tea Consumption on Cognition, Sleep, and Mood, and Understanding Individual Characteristics That Affect Responses: a Series of N-of-1 Studies
Brief Title: Understanding the Effects of Daily Tea Consumption on Attention, Sleep, and Mood, in Healthy Adults
Acronym: Reactivi-Tea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Lipton Teas and Infusions (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 67147; MA-2021-02122N (Other Grant/Funding Number: Lipton Teas and Infusions)
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: The Focus of the Study is Healthy Volunteers
Keywords: Tea; Camellia sinensis; Cognition; Mood; Sleep; Black tea; Green tea; Theanine; Caffeine; N-of-1

STUDY DESIGN:
Intervention Model Description: The study will employ an N-of-1 study design in which 30 participants will be recruited and studied over 12 weeks. In each N-of-1 study, interventions will be delivered for six days at a time, with a one day washout in between each intervention, in four blocks of three weeks, such that each intervention is received once in each three-week block. Three intervention sequences for each arm were determined by randomly selecting four out of the six possible combinations of three interventions, and ordering the four combinations so that no intervention was preceded, or followed, by itself.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Series of n-of-1 trials administering black tea interventions (Other): A series of n-of-1 trials in which participants will receive 'black tea', 'caffeine-only black tea', and 'placebo black tea'.
  Interventions: Other: Black tea flavoured, tea drink; Other: Black tea flavoured, caffeine-only drink; Other: Black tea flavoured, placebo drink
- Series of n-of-1 trials administering green tea interventions (Other): A series of n-of-1 trials in which participants will receive 'green tea', 'caffeine-only green tea', and 'placebo green tea'.
  Interventions: Other: Green tea flavoured, tea drink; Other: Green tea flavoured, caffeine-only drink; Other: Green tea flavoured, placebo drink

INTERVENTIONS:
Other: Black tea flavoured, tea drink — Black tea powder containing 50.0 mg of caffeine and 11.5 mg of theanine, to be dissolved in 200 ml boiling water.
  Arms: Series of n-of-1 trials administering black tea interventions
Other: Black tea flavoured, caffeine-only drink — 50.0 mg of caffeine in a black tea-like powder i.e., matched to the 'black tea' intervention for flavour and appearance, to be dissolved in 200 ml boiling water. Caffeine is the only biologically active ingredient in this intervention.
  Arms: Series of n-of-1 trials administering black tea interventions
Other: Black tea flavoured, placebo drink — A black tea-like powder i.e., matched to the 'black tea' intervention for flavour and appearance, containing no biologically active ingredients, to be dissolved in 200 ml boiling water.
  Arms: Series of n-of-1 trials administering black tea interventions
Other: Green tea flavoured, tea drink — Green tea powder containing 30.6 mg of caffeine and 11.1 mg of theanine, to be dissolved in 200 ml boiling water.
  Arms: Series of n-of-1 trials administering green tea interventions
Other: Green tea flavoured, caffeine-only drink — 30.6 mg of caffeine in a green tea-like powder i.e., matched to the 'green tea' intervention for flavour and appearance, to be dissolved in 200 ml boiling water. Caffeine is the only biologically active ingredient in this intervention.
  Arms: Series of n-of-1 trials administering green tea interventions
Other: Green tea flavoured, placebo drink — A green tea-like powder i.e., matched to the 'green tea' intervention for flavour and appearance, containing no biologically active ingredients, to be dissolved in 200 ml boiling water.
  Arms: Series of n-of-1 trials administering green tea interventions

SUMMARY:
The goal of these series of N-of-1 trials is to compare the effects of three tea interventions on cognition, mood, and sleep, in healthy adult participants. The main questions they aim to answer are:

* What are the short-term effects of, and differences between, three different black tea interventions on cognition, mood, and sleep, in individual participants?
* What are the short-term effects of, and differences between, three different green tea interventions on cognition, mood, and sleep, in individual participants?
* Are there any other lifestyle factors that influence the relationship between tea intake and cognition, mood, or sleep, and to what extent do they have an effect?

Participants will be asked to drink three different tea interventions in four blocks of three weeks, where each week is assigned one tea intervention. At regular intervals three times per day, seven days per week, for the 12-week study duration, participants will be asked to complete a sleep questionnaire, mood questionnaire, personalised questionnaire (with questions pertaining to physical activity and work, for example), a tea consumption recall questionnaire, and two cognitive tasks based on attention (lasting one minute each). These questionnaires and tasks comprise one measurement point and take approximately five to six minutes to complete.

DETAILED DESCRIPTION:
Two independent series of 12-week N-of-1 studies will be conducted to separately assess the effects of two primary interventions, black tea flavoured tea drink (containing bioactive compounds equivalent to naturally occurring levels in black tea), and green tea flavoured tea drink (containing bioactive compounds equivalent to naturally occurring levels in green tea), against two controls each (caffeine only, and placebo, flavoured according to the primary interventions), on cognition, mood, and sleep.

For each primary intervention, the 12-week study duration will comprise of four, three-week cycles and each cycle will comprise of three, one-week intervention periods. The order of the three interventions will be determined separately for each participant by randomly selecting four of the six possible combinations of three interventions, and such that no intervention is given in consecutive weeks. Each one-week intervention period will be split into six test days and one washout day. The washout day will be a minimum of 24 hours (00:00 to 23:59). On each of the test days, participants will be asked to drink the tea intervention allocated to that week, as often as they would like. Participants will be asked to refrain from drinking any other tea products, and caffeinated, or decaffeinated, drinks. On washout days participants will also be asked to refrain from drinking the tea products provided as part of the study.

The randomisation process to determine intervention sequences will be conducted by a third party who will not be involved in running of the study or data analysis. Each tea intervention will be coded prior to being delivered to the Rowett Institute and the file linking each tea code to the tea will be sent from Lipton Teas and Infusions to the Quality Assurance Manager for the Rowett Institute. The principal and sub-investigators will be informed which three tea codes relate to the three green tea and three black tea interventions for the purposes of running the study. The specific tea interventions assigned to each code will only be revealed to the principal and sub-investigators once the data analysis for all participants has been completed.

At three time points on each study day, participants will be prompted to complete a series of questionnaires and cognitive tasks which will form one measurement point. These time points will be decided on a per participant basis and where possible one measurement point will fall within each of the following time periods: 0800-1000, 1200-1400, 1600-1800. For participants who work night shifts these time periods will not apply, however, the time intervals between each measurement point will be maintained where possible. The cognitive tasks will be the digit vigilance task and attention switching task, and questionnaires include a sleep questionnaire, mood questionnaire, personalised questionnaire, and tea recall questionnaire. The investigators will use Gorilla Experiment Builder to deliver the questionnaires and cognitive tasks. The sleep questionnaire will only be included in the first measurement point of each day. The investigators will also ask participants to note accidental consumption of any tea or caffeine products not related to the study, but participants will not excluded from the study if they have consumed a product unrelated to the study.

Once potential participants have been screened against the inclusion and exclusion criteria and informed consent has been obtained, participants will complete a series of questionnaires that will be used to identify variables that are likely to show some degree of personal variability over time and may influence their cognition/attention, mood, sleep, and/or compliance to the intervention. Four validated questionnaires will be used: the UK Short-form 12 health questionnaire, the short-form International Physical Activity Questionnaire, the Pittsburgh Sleep Quality Index, and the trait anxiety arm of the State Trait Anxiety Inventory in order to provide an overview of their typical lifestyle-related behaviours. Participants will also be asked to complete a questionnaire detailing their tea consumption and consumption of other caffeinated food and drinks and a questionnaire to establish other lifestyle factors e.g., work routine, dependents, whether the participant lives with another person. The tea consumption questionnaire will also inform whether the participant will be included in the black tea or green tea study. Assessment of these time-dependent variables during the study is known as ecological momentary assessment and will be implemented using semi-personalised short questionnaires delivered via Gorilla Experiment Builder at each of the three daily measurement points over the course of the study.

After receiving their questionnaire responses, an in-person meeting with each participant will be arranged at a time convenient to them. This meeting will be used to determine the prompting times and to familiarise participants with the Gorilla Experiment Builder test platform, provide them with a PRO-Diary, and the tea products for the first cycle of the study.

Subsequent visits will occur every three weeks - at the end of each cycle. Participants will receive their tea products, the PRO-Diary device will be swapped with a fully charged device, and the visits will provide another opportunity for participants to ask questions or express any concerns they may have. At the end of week 12, participants will be invited to the Rowett for a final debrief and to return the PRO-Diary device.

Descriptive, univariable, and multivariable analyses will be performed in R. Owing to the personalised nature of the ecological momentary assessment and the longitudinal nature of the outcomes, individualised dynamic modelling will be the primary method of analysis for investigating both trends in variables over time, and the effect of individual-specific predictors on the attentional aspect of cognition (mean reaction times and accuracy for the attention switching task and digit vigilance task), sleep, and mood.

Individualised dynamic modelling analyses will be conducted for each participant to capture variation in the primary and secondary outcomes, and to develop unique regression models to consider the influence of individualised time-dependent predictors on the daily outcomes. Dynamic modelling includes two sets of covariates. The first set of covariates include the potential predictors exogenous to the participant (e.g., time, day of the week) and endogenous (e.g., mood, length of sleep) on the model, to identify which factors affect behaviour while controlling for the effect of time. Dynamic covariates are also included to summarise the effect of the past in present response and predictors by including lagged variables (values from previous day or two days before) of both the response and predictors, which enables us to see how much the previous state of the individuals can affect present outcomes.

ELIGIBILITY:
Inclusion Criteria:

* People that speak English
* People that possess a computer, tablet, or smartphone that they can access regularly throughout any day of the week.

Exclusion Criteria:

* A current clinical diagnosis of Alzheimer's disease
* A current clinical diagnosis of Parkinson's disease
* A current clinical diagnosis of dementia
* A current clinical diagnosis of any other brain disease
* A current clinical diagnosis of cognitive impairment
* A current clinical diagnosis of any mood disorder
* People with any food allergies
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
The cognitive domain 'attention' measured using mean reaction time and accuracy in the attention switching task | From enrolment to the end of the final tea intervention. This is the total study duration of 12 weeks.
  Participants will be presented with consecutive pairs of semi-random (a random pair from the pre-defined groups with lagged replacement, i.e., a character in one pair cannot be present in the following pair) alphanumeric characters; each pair being displayed for one second. Each pair will consist of one letter (A, E, I, U, G, K, M, R) and one number (2, 3, 4, 5, 6, 7, 8, 9), in either font colour red or purple. One character will be to the left, and one to the right, of a central fixation cross; there is equal probability of the letter or number appearing on either side. The font colour changes every three pairs. No letter or number will appear in consecutive pairs. A response is made by pressing the spacebar or tapping the screen. The two conditions for a participant to respond are: if the font colour is red and the letter is a vowel; the font colour is purple, and the number is even. In other conditions, participants should withhold from responding. The task will last one minute.
The cognitive domain 'attention' measured using mean reaction time and accuracy in the digit vigilance task | From enrolment to the end of the final tea intervention. This is the total study duration of 12 weeks.
  Participants will be shown two streams of numbers, one of the pair on the left of the screen, and one on the right. The number on the right is the target digit and the number on the left is the random digit. The target digit is a random number between 1 and 9 that is constant for the duration of the test but random at every test occasion, and the random number stream displays random numbers between 1 and 9, consecutively, for 0.75 seconds each. No two consecutive random numbers are the same. Participants should respond by pressing the spacebar on a computer, or tapping the screen on a mobile phone or tablet, as quickly as possible, when the random digit matches the target digit. The task will last one minute and a total of 15 matches will be displayed.

SECONDARY OUTCOMES:
Mood attributes measured using the Caffeine Research Visual Analogue Scale | From enrolment to the end of the final tea intervention. This is the total study duration of 12 weeks.
  The following mood outcomes are each assessed using a visual analogue scale of 0 to 100: relaxed, alert, jittery, tired, tense, headache, mentally fatigued, overall mood. Two additional mood adjectives were added: calm, energetic.
Sleep attributes measured using components of the Leeds Sleep Evaluation Questionnaire and sleep and wake times | From enrolment to the end of the final tea intervention. This is the total study duration of 12 weeks.
  All participants will be asked four questions to assess their sleep. Two are from the Leeds Sleep Evaluation Questionnaire: 'How does the way you fell asleep last night compare with how you usually fall asleep?' answered using three visual analogue scale prompts: 1. 'Harder than usual' ↔ 'Easier than usual', 2. 'Slower than usual' ↔ 'Faster than usual', 3. 'I felt less drowsy than usual' ↔ 'I felt more drowsy than usual'; 'How does your quality of sleep last night compare with your usual quality of sleep?' answered using two visual analogue scale prompts, 1. 'More restless than usual' ↔ 'Calmer than usual', 2. 'More periods of wakefulness' ↔ 'Fewer periods of wakefulness'. The other two questions concern sleep and wake times: 'What time did you turn off your light before going to sleep last night?'; 'What time did you wake up this morning?' These four questions will only be asked at the first measurement point of each test day.

CONTACTS AND LOCATIONS:
Overall Officials: Baukje d Roos, PhD, Principal Investigator — The Rowett Institute
Locations (1):
- The Rowett Institute, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No